CLINICAL TRIAL: NCT01358279
Title: Manho Kim, MD, PhD Professor, Neurology Seoul National University Hospital,
Brief Title: Transcranial Direct Current Stimulation for Migraine Attack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Manho Kim, Manho Kim, MD, PhD Professor, Neurology Seoul National University Hospital, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-4615-A
Record Dates: First submitted 2011-05-18; First posted 2011-05-23 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Acute Migraine
MeSH Terms: interventions — Transcranial Direct Current Stimulation

ARMS (1):
- migraine (Experimental)
  Interventions: Procedure: transcranial direct current stimulation

INTERVENTIONS:
Procedure: transcranial direct current stimulation — A constant current of 2 mA intensity applied for 20 min over C3 or C4

SUMMARY:
This study is conducted to investigate the therapeutic efficacy and safety of transcranial direct current stimulation (tDCS) over the primary motor cortex of patients with acute migraine attack.

ELIGIBILITY:
Inclusion Criteria:

* Aged 17-70 years
* Migraine

  * With or without aura
  * The first attack of migraine was earlier than 50 years of age
  * One to 8 moderate to severe migraine attacks per month in the 2 months preceding the screening
* Willing and able to give written informed consent
* Able to read, comprehend and complete the diary form

Exclusion Criteria:

* Not able to distinguish between migraine and non-migraine headache
* Combined headache, including the tension type headache and medication overuse headache
* Pregnant, actively trying to become pregnant or breast-feeding women
* Uncontrolled and significant medical illness
* Vertebrobasilar or hemiplegic migraine according to the International Headache Society diagnostic criteria
* Having intracranial metal implants or a cardiac pacemaker
* A history of epilepsy or other organic brain disorders
* A history of psychological diseases
* Having changed medications for migraine within 1 month before giving us informed consent
* Drug abuser or alcoholics

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-01; Primary Completion 2009-10 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Number of participants who experienced pain relief of one level or more | at 2h post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea